CLINICAL TRIAL: NCT01854372
Title: Rituximab-HyperCVAD (R-HCVAD) Alternating With Rituximab-Methotrexate-Cytarabine- (R-MC) in Newly Diagnosed Patients With Diffuse Large B-Cell Lymphoma With MYC-Rearrangement. A Phase 2, Multi-Center, Open Label Study (CTRC# 11-53)
Brief Title: Rituximab-HyperCVAD (R-HCVAD) Alternating With Rituximab-Methotrexate-Cytarabine- (R-MC) in Newly Diagnosed Patients With Diffuse Large B-Cell Lymphoma With MYC-Rearrangement.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 11-53
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Newly Diagnosed Diffuse Large B-Cell Lymphoma; Intermediate (Burkitt-Like) Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-HCVAD and R-MC Chemotherapy (Experimental): R-HCVAD - Rituximab (375 mg/m2), Cyclophosphamide (300 mg/m2), Mesna (600 mg/m2), Doxorubicin (50 mg/m2), Vincristine (2 mg total), Dexamethasone (40 mg total), Methotrexate (12 mg), Cytarabine (100mg).
  R-MC -Rituximab (375 mg/m2),Methotrexate (200 mg/m2 - 800mg/m2), Cytarabine (3000mg/m2), Leucovorin (15mg - 50mg).
  Interventions: Drug: R-HCVAD and R-MC

INTERVENTIONS:
Drug: R-HCVAD and R-MC

SUMMARY:
To estimate the I-year progression-free survival probability in patients up to 70 years of age with previously untreated diffuse large B-celllymphoma (DLBCL), or with intermediate (Burkitt-like) lymphoma, whose tumor cells show MYC rearrangement, and who are treated with alternating cycles of Rituximab-HCV AD and Rituximab-Methotrexate-Cytarabine, in concert with optimal supportive treatment including Pegfilgrastim, prophylactic antimicrobials, and close clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Diffuse large B-cell lymphoma or intermediate ("Burkitt-like") lymphoma, newly diagnosed from an excisional biopsy or from a large core biopsy with sufficient diagnostic material to perform genetic testing for MYC-R.
2. Positivity for MYC-R by Fluorescent in-situ Hybridization (FISH) or by classical cytogenetics.
3. No prior lymphoma treatment, with one exception: One cycle of R-CHOP regimen is permitted (consisting of one single dose each of Rituximab, of cyclophosphamide, of doxorubicine, and of vincristine, as well as up to 5 doses of Prednisone when part of chemotherapy).
4. No prior radiation therapy is permitted
5. Age ≥ 18 years to 70 years of age
6. CT imaging of neck, chest, abdomen and pelvis within 28 days prior to registration. Any additional imaging used to assess extent of disease must also have been done within 28 days prior to registration
7. Bidimensionally measurable disease by imaging within 28 days prior to registration
8. Adequate bone marrow biopsy, and aspiration performed for staging within 28 days before registration, and before start of any treatment
9. Indication for primary treatment with systemic multiagent chemotherapy
10. Creatinine ≤ 2.0 mg/dL and estimated (Cockroft-Gault) creatinine clearance> 50 ml/min within 7 days prior to registration
11. Cardiac ejection fraction of ≥ 50% by MUGA scan or by 2-D echocardiogram , as well as EKG without significant abnormality within 28 days prior to registration
12. Performance status of 0, of 1, or of 2 (ECOG scale)
13. Patient willing to have, and to maintain, a central venous line throughout the treatment phase (either PICC line, or double lumen tunnelled catheter, or double lumen subcutaneous venous port system)
14. Willing and logistically able to be followed as outpatient at least twice weekly, during the treatment phase.
15. Signed informed consent to accept transfusion of blood products as medically indicated
16. Signed informed consent to participate in this trial

Exclusion Criteria:

1. Age > 70 years
2. Leukemic presentation, or no evidence of disease by imaging
3. Unwilling to be screened for HIV. HIV positive patients must receive combined antiretroviral treatment while on study. They are excluded from participation unless they show a CD4 count >250/uL and a viral load < 50 within 28 days of registration.
4. Hepatic involvement and total serum bilirubin ≥ 5 mg/dL within 7 days prior to registration, or total serum bilirubin ≥ 1.6 mg/ dL without hepatic involvement within 7 days prior to registration
5. Patients with bone marrow involvement and either ANC < 1000/uLor Platelets < 50,000/uL, within 7 days before registration
6. Patients without bone marrow involvement by lymphoma, and either ANC < 1500/uL or Platelets < 100,000/uL within 7 days before registration
7. Patients with myelodysplastic syndrome, with sickle cell disease, or with transfusion dependence for over 6 months antedating the diagnosis oflymphoma.
8. Known hypersensitivity to E. coli derived proteins
9. Patients at risk of reactivation of hepatitis B who are unwilling to be treated with appropriate antivirals as medically indicated.
10. Pregnant or nursing women, or any patient with reproductive potential and unwilling to use effective contraceptive method from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method, or total abstinence.
11. Additional or prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for ~ 5 years
12. Unwilling to receive transfusions of blood products as medically indicated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival verified by PET scan. | 6 weeks